CLINICAL TRIAL: NCT01461993
Title: A Phase 2, Randomized, Active-controlled, Observer-blinded Trial, To Assess The Safety, Tolerability, And Immunogenicity Of Gardasil (Registered) (Hpv) Vaccine And Bivalent Rlp2086 Vaccine When Administered Concomitantly In Healthy Subjects Aged >=11 To <18 Years
Brief Title: A Clinical Trial to Study the Safety, Tolerance and Immunogenic Response to Gardasil and Bivalent rLP2086 Vaccine When Given at the Same Time to Children Between the Ages of 11 and 17
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Prevention
Other Study IDs: B1971011; 6108A1-2007 (Other: Alias Study Number)
Record Dates: First submitted 2011-09-28; First posted 2011-10-28 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Vaccines; Meningococcal Vaccines
Keywords: vaccine; rLP2086; Gardasil; HPV; meningitis B; N. meningitidis serogroup B; adolescents; single-blind; Meningococcal Vaccines
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; factor H-binding protein, Neisseria meningitidis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): rLP2086 + Gardasil
  Interventions: Biological: rLP2086 and Gardasil
- Group 2 (Placebo Comparator): rLP2086 and saline
  Interventions: Biological: rLP2086
- Group 3 (Active Comparator): Saline + Gardasil
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: rLP2086 and Gardasil — Gardasil vaccine and rLP2086 injection will be given to the subject concomitantly in Group 1 at Months 0, 2 and 6.
  Arms: Group 1
Biological: rLP2086 — Injections of rLP2086 and saline will be given to the subject concomitantly in Group 2 at Months 0, 2 and 6.
  Arms: Group 2
Biological: Gardasil — Injections of saline and Gardasil vaccine will be given to the subject concomitantly in Group 3 at Months 0, 2 and 6.
  Arms: Group 3

SUMMARY:
This is a clinical study to assess the safety, tolerance and immunogenic response to Gardasil (human papilloma virus (HPV)) and rLP2086 vaccine. Healthy male and female subjects will be randomized into 1 of 3 groups; the trial will be an observer-blinded study to the injection being given; and, vaccinated with either Gardasil and rLP2086 concomitantly, rLP2086 and saline concomitantly, or Gardasil and saline concomitantly. The subjects are adolescent children between the ages of 11 and 17 years old.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects from 11 to 17 years old at the time of they start the study.
* Subject must be healthy which will be determined by obtaining subject's medical history, receiving a physical examination and by judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* Previous vaccination with any HPV vaccine.
* Contraindication to vaccination with Gardasil or any HPV vaccine.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2499 (Actual)
Dates: Start 2011-09-28 (Actual); Primary Completion 2013-07-06 (Actual); Study Completion 2013-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (83):
- United States (83):
  - Coastal Clinical Research Inc., Daphne, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - The Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - West Coast Clinical Trials, LLC, Cypress, California
  - Pediatric Care Medical Group, Huntington Beach, California
  - Loma Linda University Health Care - Moreno Valley Pediatrics, Moreno Valley, California
  - Bayview Research Group, LLC, Paramount, California
  - Center for Clinical Trials, LLC, Paramount, California
  - California Research Foundation, San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Miami Research Associates, Miami, Florida
  - Pediatrics and Adolescent Medicine, PA, Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Pediatrics and Adolescent Medicine, Woodstock, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Northpoint Pediatrics, LLC, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Allina Health Bandana Square Clinic, Saint Paul, Minnesota
  - Aspen Medical Group / Odyssey Research, Saint Paul, Minnesota
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Rochester Clinical Research, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cary Pediatric Center, Cary, North Carolina
  - Duke University Medical Center - Duke Health Center, Durham, North Carolina
  - Durham Pediatrics, Durham, North Carolina
  - Duke Health Center, Durham, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Internal Medicine Consultants, Inc, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Innovis Health, LLC dba Essentia Health South University Clinic, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio
  - Senders Pediatrics, Cleveland, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Lynn Institute of Norman (LION), Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma State University - Center for Health Sciences - Pediatric Research Houston Center, Tulsa, Oklahoma
  - Oklahoma State University - Center for Health Sciences Houston Parke Physicians, Tulsa, Oklahoma
  - Preferred Primary Care Physicians, Inc., Carnegie, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Pennridge Pediatric Associates, Sellersville, Pennsylvania
  - Richard K. Ohnmacht, MD, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Charleston Pediatrics, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - The Office of Dr. Roberta Braun, MD, Austin, Texas
  - Advances In Health, Inc., Houston, Texas
  - Pediatric Healthcare of Northwest Houston, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - University of Texas Medical Branch Pediatric Specialty Center, League City, Texas
  - Benchmark Research, San Angelo, Texas
  - Clinical Trials Of Texas, Inc, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - First Steps Pediatrics, San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Pediatric Healthcare of Northwest Houston, PA, Tomball, Texas
  - Pediatric Healthcare of Northwest Houston, Tomball, Texas
  - Murray Pediatrics, Murray, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Pediatric Associates of Charlottesville, Charlottesville, Virginia
  - West Office - Pediatric Associates of Charlottesville, Charlottesville, Virginia
  - North Office - Pediatric Associates of Charlottesville, Charlottesville, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - The Vancouver Clinic, Vancouver, Washington
  - Monroe Clinic, Monroe, Wisconsin

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: rLP2086 + Gardasil; Group 2: rLP2086 + Saline; Group 3: Saline + Gardasil: Randomized to receive on a 0, 2-, 6- month schedule
Period: Overall Study
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline | Group 3: Saline + Gardasil
Started | 999 | 998 | 502
Completed | 848 | 841 | 438
Not Completed | 151 | 157 | 64
Not completed — Withdrawal by Subject | 60 | 53 | 16
Not completed — Lost to Follow-up | 44 | 48 | 22
Not completed — Protocol Violation | 10 | 9 | 7
Not completed — Adverse Event | 9 | 11 | 3
Not completed — No longer met eligibility criteria | 13 | 18 | 10
Not completed — Did not meet entrance criteria | 2 | 3 | 0
Not completed — Other | 13 | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline | Group 3: Saline + Gardasil | Total
Number analyzed (Participants) | 999 | 998 | 502 | 2499
Age, Customized [Number; unit: participants]
  11 - less than (<) 15 years | 647 | 660 | 343 | 1650
  15 - <18 years | 352 | 338 | 159 | 849
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 332 | 170 | 843
  Male | 658 | 666 | 332 | 1656

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Human Papillomavirus (HPV) Antigens
Time Frame: 1 month after Vaccination 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: rLP2086 + Gardasil | Group 3: Saline + Gardasil
Number analyzed (Participants) | 813 | 423
titer
  HPV-6 | 451.8 [417.50 to 489.01] | 550.3 [490.44 to 617.58]
  HPV-11 | 892.9 [839.52 to 949.57] | 1084.3 [997.28 to 1178.96]
  HPV-16 | 3695.4 [3426.32 to 3985.67] | 4763.4 [4285.85 to 5294.21]
  HPV-18 | 744.0 [687.67 to 804.96] | 1047.4 [939.00 to 1168.25]
Statistical Analysis 1: Comparison: Group 1: rLP2086 + Gardasil vs Group 3: Saline + Gardasil; HPV-6; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.82, 95% CI [0.72 to 0.94]
Statistical Analysis 2: Comparison: Group 1: rLP2086 + Gardasil vs Group 3: Saline + Gardasil; HPV-11; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.82, 95% CI 2-sided [0.74 to 0.91]
Statistical Analysis 3: Comparison: Group 1: rLP2086 + Gardasil vs Group 3: Saline + Gardasil; HPV-16; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.78, 95% CI 2-sided [0.68 to 0.88]
Statistical Analysis 4: Comparison: Group 1: rLP2086 + Gardasil vs Group 3: Saline + Gardasil; HPV-18; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.71, 95% CI 2-sided [0.62 to 0.81]

2. Primary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) GMTs of PMB80 [A22] and PMB2948 [B24]
Time Frame: 1 month after Vaccination 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline
Number analyzed (Participants) | 814 | 812
titer
  PMB80 [A22] (N= 803, 801) | 53.3 [50.22 to 56.66] | 57.8 [54.44 to 61.44]
  PMB2948 [B24] (N= 788, 793) | 25.8 [24.14 to 27.56] | 28.0 [26.24 to 29.87]
Statistical Analysis 1: Comparison: Group 1: rLP2086 + Gardasil vs Group 2: rLP2086 + Saline; PMB80 [A22]; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.92, 95% CI 2-sided [0.85 to 1.00]
Statistical Analysis 2: Comparison: Group 1: rLP2086 + Gardasil vs Group 2: rLP2086 + Saline; PMB2948 [B24]; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold; GMT Ratio = 0.92, 95% CI 2-sided [0.84 to 1.01]

3. Secondary Outcome: Percentage of Participants Achieving Seroconversion for Human Papillomavirus (HPV)
Time Frame: 1 month after Vaccination 3
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Gardasil | Group 3: Saline + Gardasil
Number analyzed (Participants) | 809 | 419
percentage of participants
  HPV-6 (N= 802, 414) | 99.4 | 99.3
  HPV-11 (N= 801, 417) | 99.6 | 99.5
  HPV-16 (N= 800, 413) | 99.6 | 99.5
  HPV-18 (N= 805, 418) | 99.5 | 99.0

4. Secondary Outcome: Percentage of Baseline Seropositive Participants: Group 1 and 3 Participants
Time Frame: Before vaccination 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Gardasil | Group 3: Saline + Gardasil
Number analyzed (Participants) | 814 | 423
percentage of participants
  HPV-6 | 1.4 | 2.1
  HPV-11 | 1.5 | 1.4
  HPV-16 | 1.6 | 2.4
  HPV-18 | 1.0 | 1.2

5. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ)
Time Frame: Before vaccination 1, 1 month after vaccination (Vac) 2, 3
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline
Number analyzed (Participants) | 814 | 812
percentage of participants
  Before Vaccination 1:PMB80[A22] 1:16 (N= 794, 799) | 13.7 | 16.4
  1 month after Vac 2: PMB80[A22] 1:16 (N= 794, 801) | 83.0 | 85.8
  1 month after Vac 3: PMB80[A22] 1:16 (N= 803, 801) | 94.0 | 96.3
  Before Vaccination 1:PMB2001[A56] 1:8(N= 757, 740) | 9.2 | 9.3
  1 month after Vac 2: PMB2001[A56] 1:8 (N= 790,795) | 97.5 | 98.5
  1 month after Vac 3: PMB2001[A56] 1:8 (N= 796,802) | 98.9 | 99.4
  Before Vaccination 1:PMB2948[B24] 1:8(N= 801, 793) | 5.1 | 6.9
  1 month after Vac 2: PMB2948[B24] 1:8 (N= 770,770) | 70.6 | 74.2
  1 month after Vac 3: PMB2948[B24] 1:8 (N= 788,793) | 90.5 | 92.6
  Before Vaccination 1:PMB2707[B44] 1:8(N= 806, 805) | 1.4 | 2.5
  1 month after Vac 2: PMB2707[B44] 1:8 (N= 783,776) | 54.5 | 57.1
  1 month after Vac 3: PMB2707[B44] 1:8 (N= 799,795) | 82.7 | 85.7

6. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer >= Prespecified Titer Level
Time Frame: Before Vaccination 1, 1 month after Vaccination 2, 3
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline
Number analyzed (Participants) | 814 | 812
percentage of participants
  Before Vaccination 1: PMB80 [A22] 1:4 (N=794,799) | 15.2 | 18.8
  Before Vaccination 1: PMB80 [A22] 1:8 (N=794,799) | 14.2 | 17.4
  Before Vaccination 1: PMB80 [A22] 1:32 (N=794,799) | 9.4 | 10.6
  Before Vaccination 1: PMB80 [A22] 1:64 (N=794,799) | 2.8 | 3.6
  Before Vaccination 1: PMB80[A22] 1:128 (N=794,799) | 0.5 | 0.8
  1 month after Vac 2: PMB80 [A22] 1:4 (N=794,801) | 83.8 | 86.3
  1 month after Vac 2: PMB80 [A22] 1:8 (N=794,801) | 83.2 | 86.1
  1 month after Vac 2: PMB80 [A22] 1:32 (N=794,801) | 66.9 | 69.7
  1 month after Vac 2: PMB80 [A22] 1:64 (N=794,801) | 35.9 | 35.8
  1 month after Vac 2: PMB80 [A22] 1:128 (N=794,801) | 11.0 | 13.0
  1 month after Vac 3: PMB80 [A22] 1:4 (N=803,801) | 94.3 | 96.4
  1 month after Vac 3: PMB80 [A22] 1:8 (N=803,801) | 94.3 | 96.4
  1 month after Vac 3: PMB80 [A22] 1:32 (N=803,801) | 86.3 | 87.0
  1 month after Vac 3: PMB80 [A22] 1:64 (N=803,801) | 58.0 | 61.0
  1 month after Vac 3: PMB80 [A22] 1:128 (N=803,801) | 28.1 | 31.6
  Before Vaccination 1: PMB2001[A56] 1:4 (N=757,740) | 10.4 | 10.5
  Before Vaccination 1: PMB2001[A56] 1:16(N=757,740) | 9.0 | 9.1
  Before Vaccination 1: PMB2001[A56] 1:32(N=757,740) | 8.1 | 7.7
  Before Vaccination 1: PMB2001[A56] 1:64(N=757,740) | 4.9 | 4.6
  Before Vaccination 1:PMB2001[A56] 1:128(N=757,740) | 1.7 | 1.5
  1 month after Vac 2: PMB2001 [A56] 1:4 (N=790,795) | 97.8 | 98.7
  1 month after Vac 2: PMB2001[A56] 1:16 (N=790,795) | 97.2 | 98.4
  1 month after Vac 2: PMB2001[A56] 1:32 (N=790,795) | 91.3 | 93.7
  1 month after Vac 2: PMB2001[A56] 1:64 (N=790,795) | 71.6 | 76.6
  1 month after Vac 2: PMB2001[A56] 1:128(N=790,795) | 40.4 | 41.5
  1 month after Vac 3: PMB2001 [A56] 1:4 (n=796,802) | 99.1 | 99.4
  1 month after Vac 3: PMB2001[A56] 1:16 (N=796,802) | 98.9 | 99.4
  1 month after Vac 3: PMB2001[A56] 1:32 (N=796,802) | 96.7 | 97.3
  1 month after Vac 3: PMB2001[A56] 1:64 (N=796,802) | 88.1 | 89.2
  1 month after Vac 3: PMB2001[A56] 1:128(N=796,802) | 63.6 | 67.2
  Before Vaccination 1: PMB2948[B24] 1:4 (N=801,793) | 6.1 | 8.4
  Before Vaccination 1: PMB2948[B24] 1:16(N=801,793) | 4.1 | 5.4
  Before Vaccination 1: PMB2948[B24] 1:32(N=801,793) | 1.7 | 3.0
  Before Vaccination 1: PMB2948[B24] 1:64(N=801,793) | 0.6 | 1.0
  Before Vaccination 1:PMB2948[B24] 1:128(N=801,793) | 0.1 | 0.5
  1 month after Vac 2: PMB2948 [B24] 1:4 (N=770,770) | 71.9 | 77.1
  1 month after Vac 2: PMB2948[B24] 1:16 (N=770,770) | 65.2 | 68.8
  1 month after Vac 2: PMB2948[B24] 1:32 (N=770,770) | 33.9 | 38.7
  1 month after Vac 2: PMB2948[B24] 1:64 (N=770,770) | 13.1 | 12.5
  1 month after Vac 2: PMB2948[B24] 1:128(N=770,770) | 5.3 | 5.6
  1 month after Vac 3: PMB2948 [B24] 1:4 (N=788,793) | 91.1 | 92.8
  1 month after Vac 3: PMB2948[B24] 1:16 (N=788,793) | 86.3 | 89.2
  1 month after Vac 3: PMB2948[B24] 1:32 (N=788,793) | 57.2 | 60.9
  1 month after Vac 3: PMB2948[B24] 1:64 (N=788,793) | 23.9 | 25.2
  1 month after Vac 3: PMB2948[B24] 1:128(N=788,793) | 7.6 | 8.4
  Before Vaccination 1: PMB2707[B44] 1:4 (N=806,805) | 1.7 | 3.2
  Before Vaccination 1: PMB2707[B44] 1:16(N=806,805) | 1.2 | 2.1
  Before Vaccination 1: PMB2707[B44] 1:32(N=806,805) | 0.6 | 1.4
  Before Vaccination 1: PMB2707[B44] 1:64(N=806,805) | 0.1 | 0.7
  Before Vaccination 1:PMB2707[B44] 1:128(N=806,805) | 0.0 | 0.2
  1 month after Vac 2: PMB2707 [B44] 1:4 (N=783,776) | 57.7 | 60.1
  1 month after Vac 2: PMB2707[B44] 1:16 (N=783,776) | 46.4 | 49.9
  1 month after Vac 2: PMB2707[B44] 1:32 (N=783,776) | 25.7 | 26.9
  1 month after Vac 2: PMB2707[B44] 1:64 (N=783,776) | 11.2 | 11.9
  1 month after Vac 2: PMB2707[B44] 1:128(N=783,776) | 5.0 | 5.7
  1 month after Vac 3: PMB2707 [B44] 1:4 (N=799,795) | 84.4 | 86.5
  1 month after Vac 3: PMB2707[B44] 1:16 (N=799,795) | 78.0 | 82.4
  1 month after Vac 3: PMB2707[B44] 1:32 (N=799,795) | 57.7 | 62.3
  1 month after Vac 3: PMB2707[B44] 1:64 (N=799,795) | 34.7 | 39.4
  1 month after Vac 3: PMB2707[B44] 1:128(N=799,795) | 15.1 | 18.4

7. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) Geometric Mean Titer (GMT)
Time Frame: Before Vaccination 1, 1 month after Vaccination 2, 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline
Number analyzed (Participants) | 814 | 812
titer
  Before Vaccination 1: PMB80 [A22] (N=794,799) | 9.6 [9.28 to 9.96] | 9.9 [9.58 to 10.33]
  1 month after Vac 2: PMB80 [A22] (N=794,801) | 31.9 [29.96 to 33.94] | 33.7 [31.69 to 35.85]
  Before Vaccination 1: PMB2001 [A56] (N=757,740) | 5.0 [4.78 to 5.32] | 5.0 [4.75 to 5.28]
  1 month after Vac 2: PMB2001 [A56] (N=790,795) | 70.6 [66.17 to 75.34] | 76.3 [71.93 to 80.99]
  1 month after Vac 3: PMB2001 [A56] (N=796,802) | 117.2 [110.14 to 124.76] | 128.2 [120.65 to 136.27]
  Before Vaccination 1: PMB2948 [B24] (N=801,793) | 4.3 [4.23 to 4.46] | 4.5 [4.35 to 4.65]
  1 month after Vac 2: PMB2948 [B24] (N=770,770) | 15.0 [13.88 to 16.15] | 16.3 [15.15 to 17.62]
  Before Vaccination 1: PMB2707 [B44] (N=806,805) | 4.1 [4.04 to 4.15] | 4.2 [4.10 to 4.31]
  1 month after Vac 2: PMB2707 [B44] (N=783,776) | 11.1 [10.21 to 12.01] | 11.9 [10.94 to 12.96]
  1 month after Vac 3: PMB2707 [B44] (N=799,795) | 27.2 [24.99 to 29.68] | 31.9 [29.25 to 34.82]

8. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: Vaccination 1 up to 1 month after Vaccination 3
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline | Group 3: Saline + Gardasil
Number analyzed (Participants) | 992 | 990 | 501
percentage of participants | 43.9 [40.7 to 47.0] | 41.7 [38.6 to 44.9] | 49.5 [45.0 to 54.0]

ADVERSE EVENTS:
Time Frame: AE reported from Vaccination 1 to 1 month after last administration of investigational product (bivalent rLP2086/saline/Gardasil). SAE reported from Vaccination 1 to 6 months after last of investigational product (bivalent rLP2086/saline/Gardasil)
Description: Events collected on case report form were reported.
Arm/Group | Group 1: rLP2086 + Gardasil | Group 2: rLP2086 + Saline | Group 3: Saline + Gardasil
Serious Adverse Events (participants affected / at risk) | 12/992 | 16/990 | 4/501
Other Adverse Events (participants affected / at risk) | 308/992 | 289/990 | 168/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 + Gardasil (N=992) | Group 2: rLP2086 + Saline (N=990) | Group 3: Saline + Gardasil (N=501)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nodular fasciitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Cyclothymic disorder (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Oppositional defiant disorder (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 + Gardasil (N=992) | Group 2: rLP2086 + Saline (N=990) | Group 3: Saline + Gardasil (N=501)
Vomiting (Gastrointestinal disorders) | 12 | 10 | 6
Nausea (Gastrointestinal disorders) | 15 | 6 | 2
Injection site pain (General disorders) | 50 | 43 | 21
Pyrexia (General disorders) | 15 | 11 | 5
Fatigue (General disorders) | 10 | 8 | 3
Injection site swelling (General disorders) | 11 | 8 | 2
Upper respiratory tract infection (Infections and infestations) | 49 | 53 | 29
Pharyngitis (Infections and infestations) | 20 | 36 | 9
Nasopharyngitis (Infections and infestations) | 23 | 23 | 14
Pharyngitis streptococcal (Infections and infestations) | 18 | 14 | 15
Gastroenteritis (Infections and infestations) | 23 | 11 | 8
Viral infection (Infections and infestations) | 14 | 10 | 11
Sinusitis (Infections and infestations) | 18 | 11 | 5
Gastroenteritis viral (Infections and infestations) | 9 | 8 | 8
Acute sinusitis (Infections and infestations) | 5 | 13 | 6
Otitis media (Infections and infestations) | 11 | 9 | 2
Pneumonia (Infections and infestations) | 7 | 7 | 6
Viral pharyngitis (Infections and infestations) | 2 | 6 | 8
Ligament sprain (Injury, poisoning and procedural complications) | 16 | 20 | 10
Joint injury (Injury, poisoning and procedural complications) | 12 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8 | 4
Headache (Nervous system disorders) | 50 | 38 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 16 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 23 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 13 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.